CLINICAL TRIAL: NCT04144868
Title: Normobaric Hyperoxia for Intracerebral Hemorrhage A Randomized Clinical Trial
Brief Title: Normobaric Hyperoxia for Intracerebral Hemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Jiujiang University Affiliated Hospital (Other Government)
Responsible Party: Principal Investigator, Ran Meng, Chief Physician, Head of the cerebral vein disease group. Principal Investigator, Clinical Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOTCH
Record Dates: First submitted 2019-10-22; First posted 2019-10-30 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Normobaric Hyperoxia; Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Normobaric Hyperoxia; Perihematomal Edema
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Giving high-flow mask oxygen via oxygen storage face masks (100% O2, flow rate 8 L/min, 1 hour, four times daily, and 2 L/min via nasal catheter during intermittent periods, for 7 days) or not (2 L/min via nasal catheter for 7 days) at admission.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and clinical assessors were blinded to the allocation, whereas the operators and participants were not. Neurological functional evaluations, imaging and laboratory tests were conducted by personnel blinded to the protocol of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO group (Experimental): Giving high-flow mask oxygen via oxygen storage face masks (100% O2, flow rate 8 L/min, 1 hour, four times daily, and 2 L/min via nasal catheter during intermittent periods, for 7 days) immediately at admission.
  Interventions: Device: Oxygen storage face masks and nasal catheter
- Control group (Placebo Comparator): Giving 2 L/min flow of 100% O2 via nasal catheter at admission for 24 hours daily for 7 days.
  Interventions: Device: Nasal catheter

INTERVENTIONS:
Device: Oxygen storage face masks and nasal catheter — Giving high-flow mask oxygen via oxygen storage face masks (100% O2, flow rate 8 L/min, 1 hour, four times daily, and 2 L/min via nasal catheter during intermittent periods, for 7 days) immediately at admission.
  Arms: NBO group
Device: Nasal catheter — Giving 2 L/min flow of 100% O2 via nasal catheter at admission for 24 hours daily for 7 days.
  Arms: Control group

SUMMARY:
Perihematoma edema (PHE), as the major injury for intracranial hemorrhage (ICH) involves more than the initial tissue damage induced directly by the hematoma. How to improve hypoxia in perihematoma seems to be a promising therapeutic candidate paradigm for ICH due to its pivotal role in the pathogenesis of perihematomas. Normobaric hyperoxia (NBO), supplied by a face mask (such as oxygen storage face mask) with atmosphere pressure (1ATA = 101.325 kPa, 100% O2), has been considered a safe, convenient, and promising therapy for correcting various diseases and thus garnered great attention in recent years. The previous study identified that early NBO could attenuate blood-brain barrier damage, rescue penumbra and finally improve the prognosis of ischemic stroke in patients with delayed rt-PA treatment. Therefore, given the profound effectiveness in the ischemic penumbra, we hypothesized that NBO might yield additional benefits for the ischemic-hypoxic tissues surrounding the hematoma in patients with ICH. Although many clinical trials have shown the effectiveness and safety of NBO in treating ischemic stroke, there is currently a lack of trials focusing on using NBO to treat ICH. Accordingly, we conducted a proof-of-concept, single-center, randomized controlled trial to evaluate the safety and efficacy of NBO in treating ICH patients so as to explore an innovative adjuvant therapy for ICH.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is an intractable and life-threatening stroke subtype that imposes a significant impact on people's well-being and quality of life. ICH-induced mechanical compression to the surrounding brain tissue is a major injury that increases intracranial pressure (ICP). High ICP can decrease cerebral blood flow (CBF) and influence cerebral metabolism in perihematoma and even the whole brain. Decreased aerobic metabolism and perfusion in perihematomal injury can exacerbate edema and enlarge hematoma. Moreover, secondary injury in the perihematoma, such as ischemia, oxidative stress, inflammatory response, and protease release, involves more than the initial tissue damage induced directly by the hematoma. Theoretically, low CBF and abnormal metabolism in ICH patients expose the brain tissue to the ischemic-hypoxic condition, which is similar to that in the ischemic penumbra in stroke. Therefore, the key to treating ICH is to find an approach that can rescue the perihematoma. Improving hypoxia in perihematoma seems to be a promising therapeutic candidate paradigm for ICH due to its pivotal role in the pathogenesis of perihematomas.

Normobaric hyperoxia (NBO), supplied by a face mask (such as oxygen storage face mask) with atmosphere pressure (1ATA = 101.325 kPa, 100% O2), has been considered a safe, convenient, and promising therapy for correcting various diseases and thus garnered great attention in recent years. The effectiveness of NBO on ischemic stroke (IS) has been fully identified. A plethora of studies show that NBO is capable of increasing the partial pressure of oxygen (PO2), elevating the blood flow and volume, protecting the blood-brain barrier (BBB), improving oxidative metabolism, reducing free radical damage, and even relieving inflammatory response in the penumbra. Rapid amelioration of hypoxia in brain tissue can restore brain dysfunction and improve clinical prognoses. Likewise, NBO is also regarded as a promising method for treating ICH. An animal study found that NBO for a period of 6 h per day for 3 consecutive days imposed a remarkable neuroprotective effect in rat ICH, improved neurological function, reduced brain edema, downregulated HIF-1α and VEGF expression and showed a reduction in apoptotic cells in the perihematoma. Although many clinical trials have shown the effectiveness and safety of NBO in treating ischemic stroke, there is currently a lack of trials focusing on using NBO to treat ICH. Accordingly, we conducted a proof-of-concept, single-center, randomized controlled trial to evaluate the safety and efficacy of NBO in treating ICH patients so as to explore an innovative adjuvant therapy for ICH.

ELIGIBILITY:
Inclusion criteria:

1. supratentorial hematomas confirmed by admitted cranial computed tomography (CT), with the volume ranging from 10 to 30 mL;
2. age 18-80 years;
3. National Institute of Health Stroke Scale (NIHSS) ≥ 6 and Glasgow Coma Scale (GCS) > 8 at admission;
4. onset-to-enrollment time ≤ 24 h;
5. signed informed consent.

Exclusion criteria:

1. a history of ICH, ischemic attack, brain tumor, brain trauma, and other intracranial injury or disorders;
2. pre-stroke modified ranking scales (mRS) ≥ 1;
3. life-threatening condition;
4. pre-stroke complicated with austere diseases such as cancer, heart failure, and respiratory failures;
5. severe liver and kidney disorders;
6. a history of respiratory diseases;
7. poor compliance;
8. participation in other clinical trials within the previous three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Captial Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCourt R, Gould B, Kate M, Asdaghi N, Kosior JC, Coutts S, Hill MD, Demchuk A, Jeerakathil T, Emery D, Butcher KS. Blood-brain barrier compromise does not predict perihematoma edema growth in intracerebral hemorrhage. Stroke. 2015 Apr;46(4):954-60. doi: 10.1161/STROKEAHA.114.007544. Epub 2015 Feb 19. PMID 25700288
- [Background] Ding J, Zhou D, Sui M, Meng R, Chandra A, Han J, Ding Y, Ji X. The effect of normobaric oxygen in patients with acute stroke: a systematic review and meta-analysis. Neurol Res. 2018 Jun;40(6):433-444. doi: 10.1080/01616412.2018.1454091. Epub 2018 Mar 30. PMID 29600891
- [Background] Cai L, Stevenson J, Geng X, Peng C, Ji X, Xin R, Rastogi R, Sy C, Rafols JA, Ding Y. Combining Normobaric Oxygen with Ethanol or Hypothermia Prevents Brain Damage from Thromboembolic Stroke via PKC-Akt-NOX Modulation. Mol Neurobiol. 2017 Mar;54(2):1263-1277. doi: 10.1007/s12035-016-9695-7. Epub 2016 Jan 28. PMID 26820681
- [Background] Xu Q, Fan SB, Wan YL, Liu XL, Wang L. The potential long-term neurological improvement of early hyperbaric oxygen therapy on hemorrhagic stroke in the diabetics. Diabetes Res Clin Pract. 2018 Apr;138:75-80. doi: 10.1016/j.diabres.2018.01.017. Epub 2018 Feb 3. PMID 29408705
- [Background] Shi SH, Qi ZF, Luo YM, Ji XM, Liu KJ. Normobaric oxygen treatment in acute ischemic stroke: a clinical perspective. Med Gas Res. 2016 Oct 14;6(3):147-153. doi: 10.4103/2045-9912.191360. eCollection 2016 Jul-Sep. PMID 27867482
- [Background] Liang J, Qi Z, Liu W, Wang P, Shi W, Dong W, Ji X, Luo Y, Liu KJ. Normobaric hyperoxia slows blood-brain barrier damage and expands the therapeutic time window for tissue-type plasminogen activator treatment in cerebral ischemia. Stroke. 2015 May;46(5):1344-1351. doi: 10.1161/STROKEAHA.114.008599. Epub 2015 Mar 24. PMID 25804925
- [Background] Fujiwara N, Mandeville ET, Geng X, Luo Y, Arai K, Wang X, Ji X, Singhal AB, Lo EH. Effect of normobaric oxygen therapy in a rat model of intracerebral hemorrhage. Stroke. 2011 May;42(5):1469-72. doi: 10.1161/STROKEAHA.110.593350. Epub 2011 Mar 17. PMID 21415401
- [Background] You P, Lin M, Li K, Ye X, Zheng J. Normobaric oxygen therapy inhibits HIF-1alpha and VEGF expression in perihematoma and reduces neurological function defects. Neuroreport. 2016 Mar 23;27(5):329-36. doi: 10.1097/WNR.0000000000000542. PMID 26872098
- [Result] Xu H, Li R, Duan Y, Wang J, Liu S, Zhang Y, He W, Qin X, Cao G, Yang Y, Zhuge Q, Yang J, Chen W. Quantitative assessment on blood-brain barrier permeability of acute spontaneous intracerebral hemorrhage in basal ganglia: a CT perfusion study. Neuroradiology. 2017 Jul;59(7):677-684. doi: 10.1007/s00234-017-1852-9. Epub 2017 Jun 3. PMID 28580533
- [Derived] Chen Z, Ding J, Bao B, Wu M, Cao X, Li W, Wu X, Xia Z, Xiang Y, Chen L, Liu H, Ji X, Yin X, Meng R. Normobaric hyperoxia for intracerebral hemorrhage: a randomized clinical trial. BMC Med. 2025 Dec 7;24(1):21. doi: 10.1186/s12916-025-04565-2. PMID 41353144
- [Derived] Chen Z, Ding J, Wu X, Bao B, Cao X, Wu X, Yin X, Meng R. Safety and efficacy of normobaric oxygenation on rescuing acute intracerebral hemorrhage-mediated brain damage-a protocol of randomized controlled trial. Trials. 2021 Jan 26;22(1):93. doi: 10.1186/s13063-021-05048-4. PMID 33499916

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NBO Group | Control Group
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NBO Group | Control Group | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.23 (10) | 63.71 (9.58) | 62.97 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 31 | 34 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 48 | 48 | 96
Onset-to-needle time [Mean (Standard Deviation); unit: hours] | 5.85 (4.5) | 7.91 (6.18) | 6.89 (5.48)
Hypertension [Number; unit: participants] | 36 | 29 | 65
Hyperlipidemia [Number; unit: participants] | 7 | 9 | 16
Diabetes [Number; unit: participants] | 13 | 8 | 21
Stroke [Number; unit: participants] | 12 | 7 | 19
Smoking [Number; unit: participants] | 12 | 7 | 19
Drinking [Number; unit: participants] | 15 | 15 | 30
Systolic blood pressure at admission [Mean (Standard Deviation); unit: mmHg] | 159.15 (24.58) | 158.65 (27.99) | 158.90 (26.20)
Diastolic blood pressure at admission [Mean (Standard Deviation); unit: mmHg] | 92.65 (16.05) | 89.98 (14.64) | 91.31 (15.34)
GCS score [Median (Inter-Quartile Range); unit: scores] — Glasgow Coma Scale (GCS) is a practical method for the evaluation of impairment of conscious level in response to defined stimuli, which contains three parts, including eye-opening, verbal response, and motor response (scores range from 3-15, representing deep coma to normal).
  scores | 14 [12.25 to 15] | 13 [10 to 15] | 14 [12 to 15]
NIHSS score [Median (Inter-Quartile Range); unit: scores] — The National Institute of Health Stroke Scale (NIHSS) is commonly used to evaluate neurological deficits in stroke and comprises five items in 11 fields of different neurological statuses (scores range from 0-42, representing normal to severe neurological deficits).
  scores | 10 [8 to 13] | 13 [8 to 18] | 12 [8 to 16.75]
Hematoma volume [Mean (Standard Deviation); unit: mL] | 16.77 (7.18) | 17.59 (6.98) | 17.18 (7.06)
Absolute perihematoma edema volume [Mean (Standard Deviation); unit: mL] | 24.19 (9.42) | 25.55 (10.38) | 24.87 (9.88)
Relative perihematoma edema volume [Mean (Standard Deviation); unit: ratio] | 1.53 (0.49) | 1.48 (0.28) | 1.50 (0.40)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With mRS 0-3
Description: modified Rankin Scale (mRS), an ordinal global disability scale ranging from 0 (no symptoms) to 6 (death)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
Participants | 39 | 27

2. Secondary Outcome: NIHSS Scores
Description: The NIHSS is commonly used to evaluate neurological deficits in stroke and comprises five items in 11 fields of different neurological statuses (scores range from 0-42, representing normal to severe neurological deficits).
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 9 [7 to 12] | 12 [7 to 16]

3. Secondary Outcome: NIHSS Scores
Description: as for outcome 2
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 7 [5 to 11] | 10 [5.25 to 13]

4. Secondary Outcome: NIHSS Scores
Description: as for outcome 2
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 5 [3 to 7] | 7 [4 to 9]

5. Secondary Outcome: Glasgow Coma Scale
Description: Glasgow Coma Scale is a practical method for the evaluation of impairment of conscious level in response to defined stimuli, which contains three parts, including eye-opening, verbal response, and motor response (scores range from 3-15, representing deep coma to normal).
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 15 [13 to 15] | 14 [11 to 15]

6. Secondary Outcome: Glasgow Coma Scale
Description: as for outcome 5
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 15 [14 to 15] | 15 [13 to 15]

7. Secondary Outcome: Glasgow Coma Scale
Description: as for outcome 5
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 15 [15 to 15] | 15 [14 to 15]

8. Secondary Outcome: Barthel Index
Description: Barthel Index represents functional status at follow-up time, the scores of which range from 0 (complete dependence) to 100 (complete independence) measured by several items, including feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfers, and stairs.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 80 [55 to 88.75] | 47.5 [35 to 83.75]

9. Secondary Outcome: mRS Distribution
Description: modified Rankin Scale (mRS), an ordinal global disability scale ranging from 0 (no symptoms) to 6 (death)
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 48 | 48
score on scale | 2 [1 to 3] | 3 [2 to 4]

10. Secondary Outcome: Hematoma Volume
Description: Hematoma volume in cranial CT scan, calculated by the software from United Imaging (United Imaging Healthcare Co., Ltd., Shanghai, China).
Time Frame: 3 days
Population: There were 2 patients missing imaging data in each group at 3 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 46 | 46
mL | 14.89 (6.05) | 16.8 (6.76)

11. Secondary Outcome: Hematoma Volume
Description: as for outcome 10
Time Frame: 7 days
Population: There were 3 patients in the NBO group and 4 patients in the control group missing imaging data at 7 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 45 | 44
mL | 11.14 (4.93) | 13.26 (5.32)

12. Secondary Outcome: Hematoma Volume
Description: as for outcome 10
Time Frame: 14 days
Population: There were 4 patients in the NBO group and 2 patients in the control group missing imaging data at 14 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 44 | 46
mL | 5.85 (4.02) | 6.37 (4.13)

13. Secondary Outcome: Absolute Perihematomal Edema Volume
Description: Absolute perihematomal edema in cranial CT scan, calculated by the software from United Imaging (United Imaging Healthcare Co., Ltd., Shanghai, China).
Time Frame: 3 days
Population: There were 2 patients missing imaging data in each group at 3 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 46 | 46
mL | 30.51 (10.35) | 33.51 (11.67)

14. Secondary Outcome: Absolute Perihematomal Edema Volume
Description: as for outcome 13
Time Frame: 7 days
Population: There were 3 patients in the NBO group and 4 patients in the control group missing imaging data at 7 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 45 | 44
mL | 28.43 (15.59) | 37.53 (14.61)

15. Secondary Outcome: Absolute Perihematomal Edema Volume
Description: as for outcome 13
Time Frame: 14 days
Population: There were 4 patients in the NBO group and 2 patients in the control group missing imaging data at 14 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 44 | 46
mL | 16.17 (8.36) | 20.93 (12.71)

16. Secondary Outcome: Relative Perihematomal Edema Volume
Description: The relative perihematomal edema was calculated by dividing the absolute perihematomal edema volume by the baseline hematoma volume to obtain a dimensionless ratio.
Time Frame: 3 days
Population: There were 2 patients missing imaging data in each group at 3 days.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 46 | 46
ratio | 1.99 (0.58) | 1.94 (0.46)

17. Secondary Outcome: Relative Perihematomal Edema Volume
Description: as for outcome 16
Time Frame: 7 days
Population: There were 3 patients in the NBO group and 4 patients in the control group missing imaging data at 7 days.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 45 | 44
ratio | 1.69 (0.69) | 2.18 (0.67)

18. Secondary Outcome: Relative Perihematomal Edema Volume
Description: as for outcome 16
Time Frame: 14 days
Population: There were 4 patients in the NBO group and 2 patients in the control group missing imaging data at 14 days.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | NBO Group | Control Group
Number analyzed (Participants) | 44 | 46
ratio | 0.96 (0.43) | 1.23 (0.71)

ADVERSE EVENTS:
Time Frame: From randomization to 90 days.
Description: Serious adverse events are any untoward medical occurrence meeting any of the following criteria: (1) fatal (AEs causes death); (2) life-threatening; (3) causing or prolonging hospitalization; (4) disability or organ function impairment. In addition, other adverse events include pulmonary infections, acid-base imbalances, hematoma expansion, and other complications during and after interventions that are considered to be associated with the interventions.
Arm/Group | NBO Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 12/48 | 12/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBO Group (N=48) | Control Group (N=48)
Hematoma Expansion (Vascular disorders) | 4 (4) | 3 (3)
Pulmonary Infections (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (12)
Acid-base imbalances (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT04144868/Prot_SAP_000.pdf